CLINICAL TRIAL: NCT00480753
Title: Phase II Dose Response Study of a Topical Gel Formulation of Nitroglycerin, MQX-503, in the Treatment of Raynaud's Phenomenon
Brief Title: Dose Response Study of a Topical Formulation of Nitroglycerin for the Treatment of Raynaud's Phenomenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-003
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Raynaud's Disease
Keywords: Raynaud's phenomenon; Raynaud's Disease; Raynaud's disease secondary to scleroderma; Raynaud's phenomenon secondary to autoimmune disease
MeSH Terms: conditions — Raynaud Disease | interventions — Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin

SUMMARY:
The purpose of this clinical study is to determine the response to two different dosage strengths of a topical nitroglycerin gel in patients with Raynaud's Phenomenon. Patient fingers will be monitored for changes in blood flow and skin temperature. Symptoms of pain, tingling and numbness will also be monitored.

DETAILED DESCRIPTION:
It is the intention of this protocol to study, in a controlled manner, the response of fingers of patients with Raynaud's phenomenon to two dosage strengths of a fast acting topical formulation of Nitroglycerin, MQX-503. Patients may have moderate to severe primary Raynaud's phenomenon or Raynaud's phenomenon secondary to autoimmune diseases such as scleroderma.

Quantitative changes in blood flow in the fingers of the non-dominant hand will be measured after the clinical induction of constriction of blood vessels by exposure to local cold temperatures. Secondarily, the quantitative reduction in skin temperature recovery time and symptoms of pain, tingling and numbness associated with Raynaud's phenomenon will be evaluated using a patient hand symptom analog assessment score. The frequency and severity of adverse events associated with MQX-503 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Raynaud's phenomenon
* Patients who are willing to discontinue any current therapies for Raynaud's phenomenon

Exclusion Criteria:

* The use of any medication containing nitroglycerin or known to interact with nitroglycerin
* Patients with a history of migraine or other severe headaches
* Open skin lesions or skin conditions in the area where medication is to be applied
* Pregnant or nursing women or those wishing to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Changes in blood flow in the fingers of the non-dominant hand after the induction of constriction of blood vessels by exposure to local cold temperatures. | 130 minutes

SECONDARY OUTCOMES:
Reduction in skin temperature recovery time and symptoms in the fingers of the non-dominant hand after the induction of constriction of blood vessels by exposure to local cold temperatures. | 130 minutes
Frequency and severity of adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee Shapiro, MD, Principal Investigator — The Center for Rheumatology
Locations (1):
- The Center for Rheumatology, Albany, New York, United States